CLINICAL TRIAL: NCT06648811
Title: The Effect of Kinesio Tape on Pain Management in Laparoscopic Gynecological Surgeries: A Randomized Controlled Trial
Brief Title: The Effect of Kinesio Tape on Pain Management in Laparoscopic Gynecological Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hakan Aytan, Professor, M.D., Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/912
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Gynecological Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Experimental): Kinesio tape will be applied postoperatively to the patients in this group
  Interventions: Device: Pain management after surgery
- Control group (No Intervention): These patients will only get routine postoperative management.

INTERVENTIONS:
Device: Pain management after surgery — Kinesio tapes will be applied to the patients in the study group after gynecological laparoscopic operations. The routine pain management will also be provided in these patients in addition to the kinesio tapes. Only postoperative pain management will be provided to the patients in the control group. The patients will be consisted of only the patients who will be operated laparoscopically for gynecological diseases.
  Arms: Study group

SUMMARY:
Kinesio tapes have been used in medicine to reduce pain in various situations. It is an easy applicable and effective tape. The possible affect of this tape will be assessed in patients undergoing gynecological laparoscopic surgeries.

DETAILED DESCRIPTION:
Kinesio tape is frequently used for pain palliation in medicine including orthopedics, physical therapy and rehabilitation, and dentistry. Recent studies show that it alleviates the amount of postoperative perceived pain in obstetrics and general surgery. In our study, we plan to contribute to the medical literature by studying its effect on pain palliation in patients undergoing laparoscopic gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years old female gender benign gynecologic conditions patients who underwent laparoscopic surgery patients who do not have any predisposing factors that aggreviate pain no history of malignancy no prior abdominal surgery patients who do not regularly take antiinflammatory medication patients who give permission to participate

Exclusion Criteria:

* being younger than 18 years old non-female gender having malignancies patients who underwent laparatomy patients with predisposing factors that aggrevate pain having prior abdominal surgery patients taking regular antiinflammatory medications who do not want to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Amount of perceived pain | 36 hours from the operation
  The amount of postoperative pain will be measured by using visual analogue scales (score ranges from 0 to 100 mm, higher scores indicate more pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozdemir HN, Yildiz H, Ulger G, Akay K, Guvener O, Aytan H. The effect of Kinesio tape application on postoperative pain in patients undergoing laparoscopic gynecological surgery for benign reasons: a randomized controlled study. BMC Surg. 2025 Dec 9;26(1):28. doi: 10.1186/s12893-025-03414-6. PMID 41361306